CLINICAL TRIAL: NCT03750617
Title: Randomized Trial Comparing Gastroscopy Following Web-Mediated Risk Assessment With Routine Endoscopy Screening of Colorectal Polyps
Brief Title: Web-Mediated Risk Assessment for Endoscopic Screening of Colorectal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Key Laboratory of Cancer Biology (Network)
Collaborators: Xijing Hospital (Other); Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Dake Chu, Principal Investigator, State Key Laboratory of Cancer Biology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: xjtu-20170815
Record Dates: First submitted 2018-03-27; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Colorectal Polyp
Keywords: Colorectal Polyp; Screening; Risk assessment

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pre-endoscopic screening risk assessment (Experimental)
  Interventions: Diagnostic Test: pre-endoscopic screening risk assessment
- routine screening (No Intervention)

INTERVENTIONS:
Diagnostic Test: pre-endoscopic screening risk assessment — pre-endoscopic screening risk assessment
  Arms: pre-endoscopic screening risk assessment

SUMMARY:
Colorectal polyps are risk factors for cancer. Early detection of polyps is critical for colorectal cancer management. However, the diagnosis rate of patients with colorectal polyps is still low. Therefore, we design this study to access whether pre-endoscopic screening risk assessment of genetic and environmental risk factors could improve diagnosis rate of colorectal polyps.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65.
2. Signed informed consent

Exclusion Criteria:

1. Severe back ground disease including malignancy.
2. State after gastric surgery.
3. COPD, CHF, CRF and any disease with respiratory disturbances.
4. Deviation of the nasal septum, lack of venous access at the dorsum of the hand or any other technical problem prevents gastric acid collection or base excess evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic rate of patients with polyps | 2 year
  Diagnostic rate of patients with polyps

SECONDARY OUTCOMES:
Number and characteristics of polyps detected | 2 year
  Characterization of types of polyps

CONTACTS AND LOCATIONS:
Locations (1):
- State Key laboratory of Cancer Biology, Xi'an, Shaanxi, China